CLINICAL TRIAL: NCT05811429
Title: Comparison of Aerobics and Pilates Exercises on Depression and Sleep Quality in Primigravida Females
Brief Title: Comparison of Aerobics and Pilates Exercises in Primigraivda Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0514
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Depression; Sleep Quality; Primigravida Females
Keywords: Aerobic exercises; Antenatal depression; Pilates exercises; Primigravida females; Sleep quality
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Exercise; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises (Experimental): Group A will receive aerobic exercises 2 sessions per week for 8 weeks total 16 sessions will be held.
  Interventions: Other: Aerobic exercises
- Pilates exercises (Active Comparator): Group B will receive pilates exercises 2 sessions per week for 8 weeks total 16 sessions will be held.
  Interventions: Other: Pilates exercises

INTERVENTIONS:
Other: Aerobic exercises — 16 sessions for 8 weeks ,per week 2 sessions will be given.
  Arms: Aerobic exercises
Other: Pilates exercises — 16 sessions for 8 weeks ,per week 2 sessions will be given.
  Arms: Pilates exercises

SUMMARY:
Many physical changes, as well as emotional disturbance, occur during pregnancy. In addition to external physical changes, some mental health problems such as depression, sleep and psychosis significantly increase during pregnancy. Aerobic exercises during pregnancy in primigravida females has a positive effect on depression and sleep as a primary and secondary preventive strategy.

The study will be a randomized clinical trial and Setting will be children hospital and Mehmooda hospital sheikhupura. This study will be completed in ten months and convenient sampling technique will be used. Fourty two subjects will be assigned randomly by using lottery method into two groups. Group A will receive Aerobic exercises and Group B will receive Pilate exercises. Warm up (walking) and cool down period of ten minutes will be performed by both groups. Data will be collected from all participants at baseline and after 8 weeks of treatment by using CES-D and PSQI questionnaire. After assessing the data will be analyzed by using parametric or non-parametric test by using SPSS-25.

DETAILED DESCRIPTION:
Many physical changes, as well as emotional disturbance, occur during pregnancy. In addition to external physical changes, some mental health problems such as depression, sleep and psychosis significantly increase during pregnancy. Subtle changes experienced by pregnant women can transform their ability to carry out their normal roles and may affect their quality of life, even if the pregnancy is normal. Aerobic exercises during pregnancy in primigravida females has a positive effect on depression and sleep as a primary and secondary preventive strategy. Indeed, exercise has many advantages that may make it a suitable treatment for depression in pregnancy. Pilates is considered a major exercise for improving physical, psychological, and motor functions in pregnancy. This exercise includes a series of low-pressure exercise that build strength and flexibility throughout the body.

The study will be a randomized clinical trial and will be conducted in children hospital sheikhupura and Mehmooda hospital sheikhupura. This study will be completed in time duration of ten months after the approval of synopsis and convenient sampling technique will be used. Total fourty two subjects will be assigned randomly by using lottery method into two groups. Group A will receive Aerobic exercises and Group B will receive Pilate exercises. Warm up (walking) and cool down period of ten minutes will be performed by both groups. Data will be collected from all participants at baseline and after 8 weeks of treatment by using CES-D and PSQI questionnaire. After assessing the data will be analyzed by using parametric or non-parametric test by using SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35years
* First pregnancy (primigravida)
* Single pregnancy
* Third trimester (gestational week: 26 weeks to 33 weeks)
* Depressive females (the cut off score on CES-D of 16 will be used to classify women as depressed).

Exclusion Criteria:

* Gestational diabetes
* Pregnancy Hypertension
* Placenta previa
* Any previous miscarriage history
* Medically prohibited to do exercise
* Incompetent cervix
* Polyhydramnios, Oligohydramnios

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Primigravida females
Enrollment: 38 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The Center for Epidemiologic Studies Depression Scale (CES-D Scale) | 8 weeks
  The Center for Epidemiologic Studies Depression Scale (CES-D Scale) was developed for use in studies of the epidemiology of depressive symptomatology in the general population. Its purpose differs from previous depression scales which have been used chiefly for diagnosis at clinical intake and/or evaluation of severity of illness over the course of treatment. The CES-D was designed to measure current level of depressive symptomatology, with emphasis on the affective component, depressed mood. The symptoms are among those on which a diagnosis of clinical depression is based but which may also accompany other diagnoses (including normal) to some degree. The 20-item scale used in the studies reported, possible range of scores is zero to 60, with the higher scores indicating more symptoms, weighted by frequency of occurrence during the past week
The Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) was used to measure sleep quality. This tool consists of seven areas including: subjective sleep quality, sleep latency, sleep duration, sleep efficiency (the percentage of sleeping time during the time in bed), sleep disturbances (nighttime waking), use of sleeping medications, and daytime dysfunction (distress and impaired daytime functioning). Scoring of answers was based on a scale of 0 to 3 (total score of 21). Higher scores indicate poorer sleep quality. In the present study, all participants received a score of zero for area six (the use of sleeping medications) since we did not allow students who took sleeping medication to participate

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Children Hospital, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzarino M, Kerr D, Morris ME. Pilates program design and health benefits for pregnant women: A practitioners' survey. J Bodyw Mov Ther. 2018 Apr;22(2):411-417. doi: 10.1016/j.jbmt.2017.05.015. Epub 2017 May 31. PMID 29861243
- [Background] Eastwood J, Ogbo FA, Hendry A, Noble J, Page A; Early Years Research Group (EYRG). The Impact of Antenatal Depression on Perinatal Outcomes in Australian Women. PLoS One. 2017 Jan 17;12(1):e0169907. doi: 10.1371/journal.pone.0169907. eCollection 2017. PMID 28095461
- [Background] Mindell JA, Cook RA, Nikolovski J. Sleep patterns and sleep disturbances across pregnancy. Sleep Med. 2015 Apr;16(4):483-8. doi: 10.1016/j.sleep.2014.12.006. Epub 2015 Jan 5. PMID 25666847
- [Background] Lempersz C, Noben L, van Osta G, Wassen MLH, Meershoek BPJ, Bakker P, Jacquemyn Y, Cuerva MJ, Vullings R, Westerhuis MEMH, Oei GS. Intrapartum non-invasive electrophysiological monitoring: A prospective observational study. Acta Obstet Gynecol Scand. 2020 Oct;99(10):1387-1395. doi: 10.1111/aogs.13873. Epub 2020 May 17. PMID 32306380
- [Background] Rubio-Arias JA, Marin-Cascales E, Ramos-Campo DJ, Hernandez AV, Perez-Lopez FR. Effect of exercise on sleep quality and insomnia in middle-aged women: A systematic review and meta-analysis of randomized controlled trials. Maturitas. 2017 Jun;100:49-56. doi: 10.1016/j.maturitas.2017.04.003. Epub 2017 Apr 5. PMID 28539176